CLINICAL TRIAL: NCT06720532
Title: 177Lu-PSMA-KiRi-trial
Brief Title: Kidney Function and Risk Factors in Patients with Metastatic Castration-Resistant Prostate Cancer (mCRPC) Undergoing 177Lutetium-PSMA Radioligand Therapy: a Prospective Observational Study - KiRi-Trial
Acronym: KiRi
Status: Recruiting | Type: Observational
Sponsor: Hannah Schaefer (Other)
Responsible Party: Sponsor-Investigator, Hannah Schaefer, Principal Investigator, Technical University of Munich
Organization: Technical University of Munich (Other)
Other Study IDs: 2023-402-S-KK
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Kidney Disease; Radiation Nephropathy; Metastatic Castrate Resistant Prostate Cancer (mCRPC)
Keywords: mCRPC; 177Lutetium; 177Lu-PSMA; radioligand therapy
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood and urine samples are collected from the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- mCRPC Patients with 177Lutetium-PSMA RLT: Patients diagnosed with metastatic castration-resistant prostate carcinoma (mCRPC) undergoing initial treatment with 177Lutetium-PSMA radioligand therapy at the Klinikum rechts der Isar.
  Interventions: Diagnostic Test: characterization of renal function.; Diagnostic Test: Handgrip strength test; Diagnostic Test: Questionaires

INTERVENTIONS:
Diagnostic Test: characterization of renal function. — Blood and urine sample collection
Diagnostic Test: Handgrip strength test — Assess the peak isometric strength of the hand and forearm muscles, as well as their susceptibility to fatigue.
Diagnostic Test: Questionaires — The questionnaires evaluate quality of life, psychological distress, fear of progression, frailty, pain, decision regret and treatment expectations.

SUMMARY:
The goal of this observational study is to determine the impact of 177Lutetium-Prostate Specific Membrane Antigen (PSMA) Radioligand Therapy (177Lu-PSMA-RLT) on kidney function over time. The main question it aims to answer is:

What is the absolute decline in estimated glomerular filtration rate (eGFR) in patients undergoing 177Lu-PSMA-RLT after 12 and 24 months?

Patients treated with 177Lu-PSMA-RLT will have their kidney function monitored before, during, and after therapy using routine markers like creatinine and cystatin C. Additional biomarkers and urine proteomics will be collected to identify early detection markers and risk factors for chronic kidney disease (CKD). Follow-up examinations will be conducted at regular intervals up to 5 years. The study also aims to correlate clinical risk factors and patient-reported outcomes with kidney insufficiency to assess the impact of therapy and identify vulnerable patient groups.

DETAILED DESCRIPTION:
Patients with mCRPC treated at Klinikum rechts der Isar who are newly receiving therapy with 177Lu-PSMA-RLT will be included. To ensure data quality, standard operating procedures (SOPs) will be implemented for both technical measurements and data collection. Data entered into the registry will undergo double data verification against predefined rules for range and consistency with other data fields. This ensures the accuracy and reliability of the collected data. A detailed data dictionary will be maintained, describing each variable used in the registry, including its source, coding information (e.g., TNM staging system), and normal ranges if relevant. Patient reported outcomes (PROM) of cancer related symptoms and quality of life will be collected using standardized questionnaires.

Based on the power calculation, a total of 100 patients will be included in the study. These patients will be followed up for a period of up to 5 years to ensure comprehensive data collection and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mCRPC starting 177Lu-PSMA RLT at the Klinikum rechts der Isar at the time of therapy initiation (1st cycle).

Exclusion Criteria:

* Missing or incomplete informed consent.
* age below 18 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All mCRPC patients starting with 177Lu-PSMA RLT at the Klinikum rechts der Isar
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2031-08-01 (Estimated)

PRIMARY OUTCOMES:
chronic kidney disease frequency | 2 years
  The primary objective is to determine the long term frequency of chronic kidney disease as an expression of radiation nephropathy in patients treated with 177Lu-PSMA RLT, measured by the absolute decline in eGFR.

SECONDARY OUTCOMES:
Incidence of chronic kidney disease in patients with long-term survival following 177Lu-PSMA radioligand therapy | 5 years
  Determination of the incidence of chronic kidney disease in long-term survivors following 177Lu-PSMA radioligand therapy (RLT), measured by the absolute decline in eGFR.
Identification of Clinical Risk Factors for the Development of Chronic Kidney Disease (CKD). | 2 years
  Detection of clinical risk factors that promote the development of chronic kidney disease (CKD).
Identification and Correlation of Renal Biomarkers for Early Detection of High-Risk Individuals for CKD. | 2 years
  Identification of renal biomarkers for the early detection of individuals at high risk of developing chronic kidney disease (CKD). Correlation of these biomarkers with the severity and timing of CKD onset. Measurement of established markers of glomerular injury, tubular damage, endothelial dysfunction, or functional impairment using ELISA.
Elucidating Potential Pathomechanisms of Renal Damage through established Serum Biomarkers and Urine Proteomics. | 2 years
  Deciphering potential pathomechanisms of renal damage using established serum biomarkers and urine proteomics via targeted and untargeted analyses.
Effects of 177Lu-PSMA Radioligand Therapy and its Side Effects on Patient-Reported Outcomes (PROMs). | 2 years
  Measurement of quality of life, psychological distress, fear of progression, frailty, pain, decision regret, and treatment expectations using questionnaires.
Longitudinal evaluation of potential radiation nephropathy. | 2 years
  Regular assessments of kidney function will be conducted over a period of 2 years. This will allow for the identification of the onset of kidney function impairments.

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum rechts der Isar, München, Bavaria 81675, Munich, Germany

IPD SHARING:
Plan to Share IPD: No